CLINICAL TRIAL: NCT05319730
Title: A Phase 1/2 Open-Label, Umbrella Platform Design Study of Investigational Agents With or Without Pembrolizumab (MK-3475) and/or Chemotherapy in Participants With Advanced Esophageal Cancer Previously Exposed to PD-1/PD-L1 Treatment (KEYMAKER-U06): Substudy 06B
Brief Title: A Study to Evaluate Investigational Agents With or Without Pembrolizumab (MK-3475) in Participants With Advanced Esophageal Cancer Previously Exposed to Programmed Cell Death 1 Protein (PD-1)/ Programmed Cell Death Ligand 1 (PD-L1) Treatment (MK-3475-06B)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-06B; jRCT2031220582 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); 2023-505189-26-00 (Registry Identifier: EU CT); U1111-1291-1987 (Registry Identifier: UTN); MK-3475-06B (Other: MSD); KEYMAKER-U06B (Other: MSD); 2021-005443-76 (EudraCT Number)
Record Dates: First submitted 2022-04-01; First posted 2022-04-08 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal cancer; Programmed Cell Death 1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL-1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL-2, PD-L2)
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — Paclitaxel; Irinotecan; pembrolizumab; lenvatinib; Histamine Antagonists; Histamine H2 Antagonists; Acetaminophen; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Paclitaxel or irinotecan (Active Comparator): Participants receive paclitaxel 80-100 mg/m^2 intravenously (IV) on Days 1, 8, and 15 every 28-day cycle until progressive disease (PD) or discontinuation, or irinotecan 180 mg/m^2 IV on day 1 of every 14-day cycle until PD or discontinuation.
  Interventions: Drug: Paclitaxel; Drug: Irinotecan
- Pembrolizumab + MK-4830 + paclitaxel or irinotecan (Experimental): Participants receive pembrolizumab 200 mg IV once every 3 weeks (Q3W) for up to 35 cycles (cycle=21 days) or until PD or discontinuation + MK-4830 800 mg IV Q3W up to 35 infusions + paclitaxel 80-100 mg/m^2 IV on Days 1, 8, and 15 every 28-day cycle until PD or discontinuation or irinotecan 180 mg/m^2 180 mg/m^2 on day 1 every 14-day cycle until PD or discontinuation.
  Interventions: Drug: Paclitaxel; Drug: Irinotecan; Biological: Pembrolizumab; Biological: MK-4830
- Pembrolizumab + MK-4830 + lenvatinib (Experimental): Participants receive pembrolizumab 200 mg IV Q3W up to 35 cycles (cycle=21 days) until PD or discontinuation + MK-4830 800 mg IV Q3W up to 35 infusions + lenvatinib 20 mg oral administration every day until PD or discontinuation.
  Interventions: Biological: Pembrolizumab; Biological: MK-4830; Drug: Lenvatinib
- Sacituzumab tirumotecan 4 mg/kg (Experimental): Participants will receive 4 mg/kg of sacituzumab tirumotecan via IV infusion on Days 1, 15, and 29 of each 42-day cycle until discontinuation.
  Interventions: Biological: Sacituzumab tirumotecan; Drug: Antihistamine; Drug: H2 Receptor Antagonist; Drug: Acetaminophen (or equivalent); Drug: Dexamethasone (or equivalent); Drug: Steroid Mouthwash (dexamethasone or equivalent); Drug: Supportive care measures
- Sacituzumab tirumotecan 5 mg/kg (Experimental): Participants will receive 5 mg/kg of sacituzumab tirumotecan via IV infusion on Days 1, 15, and 29 of each 42-day cycle until discontinuation.
  Interventions: Biological: Sacituzumab tirumotecan; Drug: Antihistamine; Drug: H2 Receptor Antagonist; Drug: Acetaminophen (or equivalent); Drug: Dexamethasone (or equivalent); Drug: Steroid Mouthwash (dexamethasone or equivalent); Drug: Supportive care measures

INTERVENTIONS:
Drug: Paclitaxel — 80-100 mg/m^2 IV infusion, administered on days 1, 8, and 15 of every 28-day cycle.
  Arms: Paclitaxel or irinotecan; Pembrolizumab + MK-4830 + paclitaxel or irinotecan
Drug: Irinotecan — 180 mg/m^2 IV infusion, administered on day 1 of every 14-day cycle.
  Arms: Paclitaxel or irinotecan; Pembrolizumab + MK-4830 + paclitaxel or irinotecan
Biological: Pembrolizumab — 200 mg IV infusion, administered every Q3W up to 35 infusions.
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab + MK-4830 + lenvatinib; Pembrolizumab + MK-4830 + paclitaxel or irinotecan
Biological: MK-4830 — 800 mg IV infusion, administered Q3W up to 35 infusions.
  Other Names: anti-immunoglobulin-like transcript 4 (anti-ILT4)
  Arms: Pembrolizumab + MK-4830 + lenvatinib; Pembrolizumab + MK-4830 + paclitaxel or irinotecan
Drug: Lenvatinib — 20 mg oral administration every day.
  Other Names: MK-7902; LENVIMA®
  Arms: Pembrolizumab + MK-4830 + lenvatinib
Biological: Sacituzumab tirumotecan — 4 mg/kg or 5 mg/kg IV infusion on Days 1, 15, and 29 of each 42-day cycle.
  Other Names: SKB264; MK-2870; sac-TMT
  Arms: Sacituzumab tirumotecan 4 mg/kg; Sacituzumab tirumotecan 5 mg/kg
Drug: Antihistamine — Administered per product label.
  Arms: Sacituzumab tirumotecan 4 mg/kg; Sacituzumab tirumotecan 5 mg/kg
Drug: H2 Receptor Antagonist — Administered per product label.
  Arms: Sacituzumab tirumotecan 4 mg/kg; Sacituzumab tirumotecan 5 mg/kg
Drug: Acetaminophen (or equivalent) — Administered per product label.
  Arms: Sacituzumab tirumotecan 4 mg/kg; Sacituzumab tirumotecan 5 mg/kg
Drug: Dexamethasone (or equivalent) — Administered per product label.
  Arms: Sacituzumab tirumotecan 4 mg/kg; Sacituzumab tirumotecan 5 mg/kg
Drug: Steroid Mouthwash (dexamethasone or equivalent) — Administered per product label.
  Arms: Sacituzumab tirumotecan 4 mg/kg; Sacituzumab tirumotecan 5 mg/kg
Drug: Supportive care measures — Participants are allowed to take supportive care measures for the management of adverse events associated with study intervention at the discretion of the investigator. Artificial tear drops or ointment may be given as a supportive care for Ocular Surface Toxicity.
  Arms: Sacituzumab tirumotecan 4 mg/kg; Sacituzumab tirumotecan 5 mg/kg

SUMMARY:
This is a Phase 1/2, multicenter, randomized, open-label umbrella platform study to evaluate the safety and efficacy of investigational agents with or without pembrolizumab and/or chemotherapy, for the treatment of participants with second line (2L) esophageal squamous cell carcinoma (ESCC) who have previously been exposed to PD-1/PD-L1 based treatment.

DETAILED DESCRIPTION:
The master protocol is MK-3475-U06.

As of Protocol Amendment 5, the Pembrolizumab Plus MK-4830 Plus Paclitaxel/Irinotecan arm and the Pembrolizumab Plus MK-4830 Plus Lenvatinib arm are no longer actively enrolling participants.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of metastatic or locally advanced unresectable esophageal squamous cell carcinoma (ESCC)
* Has experienced investigator documented radiographic or clinical disease progression on one prior line of standard therapy, that includes a platinum agent and previous exposure to an anti-programmed cell death 1 (PD1)/programmed cell death ligand 1 (PD-L1) based immune oncology (IO) therapy
* Has provided an archival or most recent tumor tissue sample obtained as part of clinical practice
* Participants who have adverse events (AEs) due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline. Participants with endocrine-related AEs who are adequately treated with hormone replacement or participants who have ≤Grade 2 neuropathy are eligible

Exclusion Criteria:

* Direct invasion into adjacent organs such as the aorta or trachea
* Has experienced weight loss >10% over approximately 2 months prior to first dose of study therapy
* Has history of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or severe corneal disease that prevents/delays corneal healing
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous history of inflammatory bowel disease
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
* Known additional malignancy that is progressing or has required active treatment within the past 3 years, except basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ that has undergone potentially curative therapy
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Participants with human immunodeficiency virus (HIV) with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* History of allogenic tissue/solid organ transplant
* Clinically significant cardiovascular disease within 12 months from first dose of study intervention
* Has risk for significant gastrointestinal (GI) bleeding such as a serious nonhealing wound, peptic ulcer, or bone fracture within 28 days prior to allocation/randomization, significant bleeding disorders, vasculitis, or has had a significant bleeding episode from the GI tract within 12 weeks prior to allocation/randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2026-11-07 (Estimated); Study Completion 2029-04-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose-Limiting Toxicities (DLTs) During Safety Lead-in Phase | Up to approximately 3 weeks
  A DLT is defined as any drug-related AE according to the National Cancer Institute Common Terminology for Adverse Events (NCI CTCAE) Version 5.0, observed during the DLT evaluation period that results in a change to a given dose or a delay in initiating the next cycle.
Number of Participants Who Experienced an Adverse Event (AE) During Safety Lead-in Phase | Up to approximately 3 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Who Discontinue Study Treatment Due to an AE During Safety Lead-in Phase | Up to approximately 3 weeks
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE will be presented.
Objective Response Rate (ORR) | Up to approximately 41 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 70 months
  PFS is defined as the time from allocation to the first documented progressive disease (PD) as assessed by RECIST 1.1 or death due to any cause, whichever occurs first. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be presented.
Duration of Response (DOR) | Up to approximately 70 months
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Overall Survival (OS) | Up to approximately 70 months
  OS is defined as the time from the date of allocation to death from any cause.
Number of Participants Experiencing at Least One Adverse Event (AE) During the Efficacy Phase | Up to approximately 70 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Number of Participants Who Discontinue Study Treatment Due to An AE During the Efficacy Phase | Up to approximately 70 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (57):
- United States (5):
  - University of Arizona Cancer Center-University of Arizona Cancer Center ( Site 4927), Tucson, Arizona
  - UCLA Hematology/Oncology - Santa Monica ( Site 4905), Los Angeles, California
  - Hematology-Oncology Associates of Central NY, P.C. ( Site 4925), East Syracuse, New York
  - Columbia University Irving Medical Center-CUIMC Herbert Irving Comprehensive Cancer Center Clinical ( Site 4907), New York, New York
  - UPMC Hillman Cancer Center-UPMC ( Site 4904), Pittsburgh, Pennsylvania
- Brazil (3):
  - Liga Norte Riograndense Contra o Câncer ( Site 4303), Natal, Rio Grande do Norte
  - Hospital Nossa Senhora da Conceição ( Site 4301), Porto Alegre, Rio Grande do Sul
  - ICESP - INSTITUTO DO CÂNCER DO ESTADO DE SÃO PAULO ( Site 4300), São Paulo
- Chile (4):
  - FALP-UIDO ( Site 4400), Santiago, Region M. de Santiago
  - Centro de Oncología de Precisión-Oncology ( Site 4404), Santiago, Region M. de Santiago
  - Clínica las Condes ( Site 4403), Santiago, Region M. de Santiago
  - Clínica UC San Carlos de Apoquindo ( Site 4405), Santiago, Region M. de Santiago
- China (6):
  - Anhui Provincial Hospital South District ( Site 3501), Hefei, Anhui
  - Beijing Cancer hospital-Digestive Oncology ( Site 3500), Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xinxiang Medical University-Oncology ( Site 3510), Xinxiang, Henan
  - First Huai'an Hospital Affiliated to Nanjing Medical University ( Site 3506), Huai'an, Jiangsu
  - Shanghai Chest Hospital-Esophageal surgery department ( Site 3513), Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital-Thoracic oncology ( Site 3511), Hangzhou, Zhejiang
- Germany (5):
  - Institut für Klinisch Onkologische Forschung-Klink für Onkologie und Hämatologie ( Site 4801), Frankfurt am Main, Hesse
  - Universitaetsklinikum Duesseldorf ( Site 4802), Düsseldorf, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden-Medical Dept I - Medical Oncology ( Site 4806), Dresden, Saxony
  - Charité Campus Virchow-Klinikum-Klinik Hämatologie Onkologie Tumorimmunologie ( Site 4804), Berlin
  - Facharztzentrum Eppendorf ( Site 4807), Hamburg
- Italy (6):
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori"-Oncologia Medica ( Site 3207), Meldola, Emilia-Romagna
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 3200), Milan, Lombardy
  - Azienda Ospedaliero Universitaria Pisana ( Site 3206), Pisa, Tuscany
  - Istituto Oncologico Veneto IRCCS-Oncologia Medica 1 ( Site 3203), Padua, Veneto
  - Ospedale San Raffaele-Oncologia Medica ( Site 3202), Milan
  - Istituto Europeo di Oncologia IRCCS-Divisione di Sviluppo di Nuovi Farmaci per Terapie Innovative ( Site 3201), Milan
- Japan (5):
  - Aichi Cancer Center ( Site 3702), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 3701), Kashiwa, Chiba
  - Saitama Prefectural Cancer Center ( Site 3703), Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center ( Site 3704), Nagaizumi-cho,Sunto-gun, Shizuoka
  - National Cancer Center Hospital ( Site 3700), Chuo-ku, Tokyo
- Oslo universitetssykehus, Radiumhospitalet ( Site 4501), Oslo, Norway
- National University Hospital ( Site 3800), Singapore, South West, Singapore
- South Korea (2):
  - Asan Medical Center-Department of Oncology ( Site 3901), Seoul
  - Samsung Medical Center-Division of Hematology/Oncology ( Site 3900), Seoul
- Switzerland (2):
  - Hôpitaux Universitaires de Genève (HUG) ( Site 4702), Geneva, Canton of Geneva
  - Kantonsspital Graubünden-Medizin ( Site 4700), Chur, Kanton Graubünden
- Taiwan (7):
  - Chang Gung Memorial Hospital at Kaohsiung ( Site 4003), Kaohsiung Niao Sung Dist, Kaohsiung
  - China Medical University Hospital ( Site 4007), Taichung
  - Taichung Veterans General Hospital-Radiation Oncology ( Site 4008), Taichung
  - National Cheng Kung University Hospital ( Site 4001), Tainan
  - National Taiwan University Hospital ( Site 4000), Taipei
  - Taipei Veterans General Hospital ( Site 4005), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 4006), Taoyuan District
- Thailand (3):
  - Chulalongkorn University ( Site 4104), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital ( Site 4102), Bangkok, Bangkok
  - Songklanagarind hospital ( Site 4105), Hat Yai, Changwat Songkhla
- Turkey (Türkiye) (7):
  - Adana Medical Park Seyhan Hastanesi-Medikal Onkoloji ( Site 3417), Adana
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 3402), Ankara
  - Memorial Ankara Hastanesi-Medical Oncology ( Site 3408), Ankara
  - Ankara Bilkent City Hospital-Medical Oncology ( Site 3405), Ankara
  - Atatürk Üniversitesi-onkoloji ( Site 3416), Erzurum
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 3403), Istanbul
  - I.E.U. Medical Point Hastanesi-Oncology ( Site 3406), Izmir

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26275&tenant=MT_MSD_9011